CLINICAL TRIAL: NCT07330076
Title: Protocol for a Prospective, Single-arm, Multicenter Clinical Study on the Efficacy and Safety of Iruplinalkib Tablets as Postoperative Adjuvant Therapy in Stage IA ALK-positive NSCLC With High-risk Factors
Brief Title: Iruplinalkib Tablets as Postoperative Adjuvant Therapy in Stage IA ALK-positive NSCLC With High-risk Factors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20251139
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: NSCLC
Keywords: Iruplinalkib Tablets；ALK-positive；NSCLC； high-risk factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iruplinalkib Tablets (Experimental)
  Interventions: Drug: Iruplinalkib tablets

INTERVENTIONS:
Drug: Iruplinalkib tablets — Iruplinalkib: Refer to the drug insert. The tablets should be swallowed whole and must not be crushed, divided, or chewed. The recommended dosage is once daily, which can be taken on an empty stomach or with food. From Day 1 to Day 7, the dose is 60mg per administration. If tolerated, the dose should be increased to 180mg per administration starting from Day 8, and continued until disease progression, intolerable toxicity, or completion of the 2-year treatment period.If a subject misses a scheduled dose, it should be taken within 8 hours of the missed time; doses missed by more than 8 hours should not be made up. If vomiting occurs after taking a dose, no additional dose should be taken. The investigator will assess whether to continue with the next scheduled dose.

SUMMARY:
The primary objective is to evaluate the efficacy and safety of Iruplinalkib Tablets as postoperative adjuvant therapy in patients with stage IA, ALK-positive NSCLC with high-risk factors.

DETAILED DESCRIPTION:
This Prospective, Single-arm, Multicenter Clinical Study aims to evaluate the Efficacy and Safety of Iruplinalkib Tablets as Postoperative Adjuvant Therapy in Stage IA ALK-positive NSCLC with High-risk Factors.This study consists of three phases: screening, treatment, and follow-up.Efficacy evaluation and safety monitoring should be performed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

- 1.Age ≥18 years, male or female. 2.ECOG Performance Status (PS) score: 0-1. 3.Expected survival ≥12 weeks. 4.Histologically or cytologically confirmed non-small cell lung cancer. 5.ALK-positive status confirmed by the investigator (NGS). 6.Clinical stage IA (maximum tumor diameter ≤3 cm, AJCC 9th edition). 7.No prior treatment with any ALK TKI targeted therapy. 8.The patient has undergone curative-intent tumor resection (sublobar resection, lobectomy, sleeve resection).

9.Organ function meets the following requirements (use of any blood products or hematopoietic growth factors within 14 days prior to enrollment is not allowed):

* Hemoglobin ≥90 g/L;
* White blood cell count ≥3.5 × 10⁹/L;
* Absolute neutrophil count ≥1.5 × 10⁹/L;
* Platelets ≥80 × 10⁹/L;
* AST, ALT ≤2.5 × ULN; if liver metastases are present, AST, ALT ≤5 × ULN;
* Total bilirubin (TBIL) ≤1.5 × ULN;
* Urea/BUN and creatinine (Cr) ≤1.5 × ULN (and creatinine clearance (CCr) ≥50 mL/min);
* Left ventricular ejection fraction (LVEF) ≥50%. 10.Patients of childbearing potential/fertile males must agree to use effective contraception.

Exclusion Criteria:

* 1.Presence of pathological components other than non-small cell carcinoma in tissue or cytology.

  2. History of allergy to ALK TKI agents or their ingredients. 3. Poorly controlled underlying diseases before enrollment, such as coronary artery disease, heart failure, cerebral infarction, hypertension, chronic obstructive pulmonary disease, interstitial lung disease, rheumatic diseases, peptic ulcer, etc. (to be determined by the investigator's assessment).

  4. Active pulmonary tuberculosis (TB), active tuberculosis infection, or active syphilis infection; eligibility for the clinical trial may be reassessed after the condition is stably controlled.

  5. Positive anti-HIV test; positive hepatitis B surface antigen (HBsAg) with HBV-DNA above the upper limit of normal; active hepatitis C virus (HCV) infection.

  6. Serious infection within 4 weeks prior to the first dose, including but not limited to comorbidities requiring hospitalization, sepsis, or severe pneumonia; active infection requiring systemic anti-infective therapy within 2 weeks prior to the first dose (excluding antiviral therapy for hepatitis B or C).

  7. Psychiatric disorders or social conditions that limit the subject's compliance with study requirements or affect their ability to provide written informed consent.

  8. Any arterial thromboembolic event within 6 months prior to the first dose, venous thromboembolic events of Grade 3 or above, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy within 3 months prior to the first dose.

  9. History of severe bleeding tendency or coagulation dysfunction; obvious active bleeding within 1 month prior to the first dose (to be determined by the investigator's assessment).

  10. History of drug abuse, alcohol abuse, or substance abuse. 11. Pregnant or lactating women. 12. Patients deemed unsuitable for participation in this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-01-06 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year DFS rate | Up to 36 months
  Defined as the proportion of patients who have not experienced disease progression or death from any cause from the initiation of Iruplinalkib treatment until the end of the third year.

SECONDARY OUTCOMES:
Overall Survival (OS) | Time Frame: up to 36 month
  The time from the start of treatment until death.

CONTACTS AND LOCATIONS:
Overall Officials: zhenfa Zhang, M.D, Principal Investigator — Department of lung cancer, Tianjin Medical University Cancer Institute and Hospital